CLINICAL TRIAL: NCT01915134
Title: A Prospective,Randomized,Controlled,Multicenter,Phase III Study of Stage Ⅲ Study of Gemcitabine Plus Cisplatin With or Without Endostatin to the Metastatic Nasopharyngeal Carcinoma
Brief Title: Endostatin in Combination With Chemotherapy for Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejaingCH-npc-03
Record Dates: First submitted 2013-07-21; First posted 2013-08-02 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2013-07

CONDITIONS: Effects of Chemotherapy; Stage IVC Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Recombinant Human Endostatin; chemotherapy; gemcitabine and cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endostatins; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGP group (Experimental): the group of participants who undergoing Recombinant Human Endostatin plus Gemcitabine and cisplatin chemotherapy
  Interventions: Drug: Recombinant Human Endostatin plus gemcitabine and cisplatin
- GP group (Active Comparator): the group of participants who undergoing only Gemcitabine and cisplatin chemotherapy
  Interventions: Drug: Gemcitabine and cisplatin

INTERVENTIONS:
Drug: Recombinant Human Endostatin plus gemcitabine and cisplatin — target therapy plus chemotherapy:4-6 cycles of Recombinant Human Endostatin plus gemcitabine and cisplatin:Endostatin：7.5mg/m2/d,d1-14,concomitant with chemotherapy for 4-6 cycles.Gemcitabine and cisplatin:4-6 cycles of GP chemotherapy with gemcitabine 1000mg/m2,d1,8,cisplatin80mg/m2,d1.Chemotherapy will be given once every three weeks.
  Other Names: Experimental: EGP group
  Arms: EGP group
Drug: Gemcitabine and cisplatin — only chemotherapy：Gemcitabine and cisplatin:4-6 cycles of GP chemotherapy with gemcitabine 1000mg/m2,d1,8,cisplatin80mg/m2,d1.Chemotherapy will be given once every three weeks.
  Other Names: No Intervention: GP group
  Arms: GP group

SUMMARY:
The investigators designed this study to evaluate the efficiency and the acute toxicities of recombinant human endostatin (endostar) combined with chemotherapy in the metastatic nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
To evaluate the progression free survival (PFS), overall survival (OS), Acute adverse reaction of recombinant human endostatin (endostar) combined with chemotherapy to the metastatic nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* metastatic nasopharyngeal carcinoma 6 months after first treatment,never receive any anticancer treatment except local radiotherapy to the bone metastasis，at least one measurable metastatic lesions，ECOG PS 0-1，Electrocardiogram (ecg) no special abnormal，comply with the test requirements, cooperate with regular follow-up.

Exclusion Criteria:

* To give local treatment,clinical severe infection(>grade 2),with the central nervous system metastases,ECOG PS≥2,patients with pregnancy or breastfeeding,has a history of peripheral nerve disease,concomitant with other serious diseases,ever or concomitant with other serious diseases except for Cervical carcinoma in situ,cure of basal cell carcinoma,bladder surface tumor,any cancer 3 years after curation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
progress free survival(PFS) | 2years after the inception assignment
  PFS means assignment to the date of any local or distant progress of the disease using Kaplan-Meier calculate the progress free survival rates,and find out is there significant difference between these two groups.

SECONDARY OUTCOMES:
overall survival(OS) | 1 year ,2 years and 3 years after the inception of the assignment
  the overall survival denote to assignment to date of death from any cause. Using Kaplan-Meier to calculate the 2-year ,3-year,5-year overall survival rate,and find is there any significant difference between these two groups.
Adverse events | participants will be followed for the duration of hospital stay,an expected average of 100 days and every 3 months thereafter for 3 years
  observe and record the toxicity profile(including but not limit to mucositis,liver and kidney function,et al.)according NCI-CTCAE(3rd edition) during the neoadjuvant chemotherapy ,chemoradiation and follow-up.

OTHER OUTCOMES:
The quality of life assessment | participants will be followed for the duration of hospital stay,an expected average of 100 days and every 6 months thereafter for 3 years
  According to the most commonly used questionnaire EORTC QLQ C30 and H&N35 35 for evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, Principal Investigator — Zhejiang Cancer Hospital; Xiaozhong Chen, Principal Investigator — Zhejiang Cancer Hospital Hangzhou, Zhejiang, China 310022
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China